CLINICAL TRIAL: NCT04922229
Title: Comparative Effectiveness in the Management of Irreversible Pulpitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ashraf Fouad, Professor and Chair, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001234
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Irreversible Pulpitis
Keywords: Pulpotomy; Vital Pulp Therapy
MeSH Terms: interventions — Dental Implantation, Endosseous, Endodontic; Pulpotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Root canal treatment (RCT) (Active Comparator): For cases with this diagnosis RCT is the standard of care and will be done according to clinically approved protocols
  Interventions: Procedure: RCT
- Pulpotomy (Experimental): Pulpotomy with tricalcium silicates has shown high clinical success in these cases. However, it is not known how this success compares to RCT under similar conditions and with an intent-to-treat study design, which will be employed here.
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: RCT — This is the standard of care for this diagnosis
  Other Names: Endodontic therapy
  Arms: Root canal treatment (RCT)
Procedure: Pulpotomy — For cases with normal apical tissues, pulpotomy using tricalcium silicates has been shown to have high clinical success. Either partial or complete pulpotomy will be performed depending on the size of pulp exposure.
  Other Names: Therapeutic pulpotomy
  Arms: Pulpotomy

SUMMARY:
This project addresses a central question within the practice of dentistry: Is a pulpotomy procedure effective in the treatment of a tooth with symptomatic irreversible pulpitis and normal periapex? In addition, the project seeks to identify clinical and molecular biomarkers that are predictive of the success of pulpotomy.

DETAILED DESCRIPTION:
In this study, patients will be randomized to two groups. All patients will have a diagnosis of irreversible pulpitis with normal apical tissues. The groups will be root canal treatment and pulpotomy. The patients will be followed clinically and radiographically for 2 years following the treatment. Predictors of the outcome of pulpotomy will be clinical and laboratory-based parameters.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary or mandibular first or second mature permanent molars with carious lesions or restorations (excluding crowns), with signs and symptoms of symptomatic irreversible pulpitis (defined as spontaneous pulpal pain and cold hyperalgesia >30 seconds), and normal apical tissues.
* Tooth is responsive to cold and electrical pulp testing.
* Patients aged ≥12 years for first molars and ≥16 years for second molars.

Exclusion Criteria:

* Evidence of Pulp Necrosis or Apical Periodontitis, preoperatively or upon inspection of an exposure site
* Teeth that are badly broken down and/or are not restorable.
* Teeth with mechanical allodynia assessed by registering bite force that is at least 50N lower than the contralateral side.
* Teeth with radiographic evidence of internal, or external cervical, inflammatory or replacement root resorption, or with complete pulp canal obliteration.
* Radiographic evidence of PDL space wider than three times normal width
* Clinical evidence of swelling or sinus tract
* Periodontal pocket probing depth ≥5 mm in any site around the tooth.
* Clinical evidence of cracks connecting mesial and distal surfaces and/or extending in pulp chamber or associated with periodontal pockets ≥ 5 mm.
* History of taking centrally acting drugs (e.g., tricyclic antidepressants), which interfere with the release of pain mediators and/or modify pain experience, within the previous 6 months.
* Use of medications that affect the host response such as methotrexate, corticosteroids or cyclosporin.
* Patients on immunosuppressive agents, chronic corticosteroid use, autoimmune disease, or other immunocompromising diseases or medications.
* Patients who require IV sedation or general anesthesia for their dental treatment.
* Teeth with full coverage crowns.
* Teeth undergoing active orthodontic movement.
* Teeth that require elective RCTx to place a post for restorative purposes.
* Teeth with no contralateral molars with normal pulp and periapical tissues for bite and pulp testing controls.
* Teeth in the pulpotomy group in which, following complete pulpotomy, bleeding does not stop after 10 minutes with 3-4% hypochlorite cotton pellet. These will be considered treatment failure and treated with RCTx.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 138 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a successful outcome of pulpotomy versus RCT | From baseline through 2 years
  A composite of clinical and radiographic findings and incidence of follow up procedures

SECONDARY OUTCOMES:
Determine prognostic validity of preoperative hyperalgesia in determining the outcome of pulpotomy | From baseline to two years
  Neurosensory measurements of preoperative signs and symptoms will be measured and correlated with the outcome of pulpotomy
Determine prognostic validity of a set of pulpal inflammatory proteins in determining the outcome of pulpotomy | From baseline to 2 years
  Protein analysis at the time of treatment will be correlated with the outcome of pulpotomy

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Fouad, DDS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- School of Dentistry, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined